CLINICAL TRIAL: NCT01442194
Title: Long-term, Prospective,Multinational, Parallel-cohort Study Monitoring Safety in Patients With MS Newly Started With Fingolimod Once Daily or Treated With Another Approved Disease-modifying Therapy
Brief Title: Safety Study in Patients With Multiple Sclerosis Treated Fingolimod or Other Approved Disease-modifying Therapies
Acronym: PASSAGE
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CFTY720D2403
Record Dates: First submitted 2011-08-21; First posted 2011-09-28 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; fingolimod; observational study
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Fingolimod: non-interventional
  Interventions: Drug: Fingolimod
- parallel cohort: non-interventional
  Interventions: Drug: other disease-modifying therapy

INTERVENTIONS:
Drug: other disease-modifying therapy
  Groups: parallel cohort
Drug: Fingolimod
  Groups: Fingolimod

SUMMARY:
The purpose of this world-wide prospective parallel-cohort study in patients with relapsing forms of MS, either newly treated with fingolimod or receiving another disease-modifying therapy, is to further explore the incidence of selected safety- related outcomes and to further monitor the overall safety profile of fingolimod under conditions of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients that as part of their routine clinical care and according to the locally approved label, are either;
* Starting fingolimod at time of study entry.
* Starting another approved DMT or started within maximum 6 months prior to study entry.
* Patients, or a able legal representative of the patient, who are willing to provide written informed consent.

Fingolimod patients will constitute the fingolimod cohort while patients with the other DMT will constitute the parallel cohort

Exclusion Criteria:

* Patients previously or currently treated with a cytotoxic agent (e.g. mitoxantrone, cladribine, alemtuzumab) or natalizumab
* Patients participating simultaneously in another study with inclusion/exclusion criteria more restrictive than the label or an interventional study unless this is a study on fingolimod lasting 1 month maximum

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsing forms of MS that have been recently initiated on fingolimod by their treating physician or patients that are treated with other disease-modifying therapies as part of their MS treatment in accordance with the respective local prescribing information and routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 3076 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
For each of the selected safety outcomes, number of patients with a reported event since study start | Patients will be followed for an expected average of 5 years
  Incidence of AEs for bradyarrhythmias, liver toxicity, macular edema, infections

SECONDARY OUTCOMES:
Number of patients SAEs since study start | Patients will be followed for an expected average of 5 years
PRIMUS activities, comparison of mean change between the 2 cohorts | Patients will be followed for an expected average of 5 years
TSQM-9, comparison between the 2 cohorts | Patients will be followed for an expected average of 5 years
WPAI-GH, comparison of mean change between the 2 cohorts | Patients will be followed for an expected average of 5 years
MSIS-29, comparison of mean change between the 2 cohorts | Patients will be followed for an expected average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (211):
- United States (184):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Sottsdale, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Banning, California
  - Novartis Investigative Site, Burbank, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Placentia, California
  - Novartis Investigative Site, Pomona, California
  - Novartis Investigative Site, Redding, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Temecula, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Basalt, Colorado
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Louisville, Colorado
  - Novartis Investigative Site, Parker, Colorado
  - Novartis Investigative Site, Fairfield, Connecticut
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Waterbury, Connecticut
  - Novartis Investigative Site, Dover, Delaware
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Clermont, Florida
  - Novartis Investigative Site, Delray Beach, Florida
  - Novartis Investigative Site, Doral, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Naples, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Panama City, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Wellington, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Weston, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Suwanee, Georgia
  - Novartis Investigative Site, Arlington Heights, Illinois
  - Novartis Investigative Site, Carbondale, Illinois
  - Novartis Investigative Site, Flossmoor, Illinois
  - Novartis Investigative Site, Marywood, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Anderson, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Lafayette, Indiana
  - Novartis Investigative Site, Merrillville, Indiana
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Hammond, Louisiana
  - Novartis Investigative Site, Auburn, Maine
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Bethesda, Maryland
  - Novartis Investigative Site, Charlotte Hall, Maryland
  - Novartis Investigative Site, Hagerstown, Maryland
  - Novartis Investigative Site, Lutherville, Maryland
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Foxborough, Massachusetts
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Wellesley, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Caro, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Jackson, Michigan
  - Novartis Investigative Site, Owosso, Michigan
  - Novartis Investigative Site, Rochester Hills, Michigan
  - Novartis Investigative Site, Southfield, Michigan
  - Novartis Investigative Site, Traverse City, Michigan
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Golden Valley, Minnesota
  - Novartis Investigative Site, City of Saint Peters, Missouri
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Hastings, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Fair Lawn, New Jersey
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, Somerset, New Jersey
  - Novartis Investigative Site, West Long Branch, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Amherst, New York
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Cedarhurst, New York
  - Novartis Investigative Site, Johnson City, New York
  - Novartis Investigative Site, Kingston, New York
  - Novartis Investigative Site, Lake Success, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Patchogue, New York
  - Novartis Investigative Site, Plainview, New York
  - Novartis Investigative Site, Poughkeepsie, New York
  - Novartis Investigative Site, Staten Island, New York
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Sanford, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Bismarck, North Dakota
  - Novartis Investigative Site, Bellevue, Ohio
  - Novartis Investigative Site, Centerville, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Springfield, Oregon
  - Novartis Investigative Site, Greensburg, Pennsylvania
  - Novartis Investigative Site, Meadowbrook, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Willow Grove, Pennsylvania
  - Novartis Investigative Site, Beaufort, South Carolina
  - Novartis Investigative Site, Camden, South Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Old Point Station, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Brownwood, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Kingwood, Texas
  - Novartis Investigative Site, Mansfield, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Stafford, Texas
  - Novartis Investigative Site, Sugar Land, Texas
  - Novartis Investigative Site, Provo, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Alexandria, Virginia
  - Novartis Investigative Site, Arlington, Virginia
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, McLean, Virginia
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Vienna, Virginia
  - Novartis Investigative Site, Winchester, Virginia
  - Novartis Investigative Site, Richland, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Wenatchee, Washington
  - Novartis Investigative Site, Beckley, West Virginia
  - Novartis Investigative Site, Huntington, West Virginia
  - Novartis Investigative Site, Green Bay, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
  - Novartis Investigative Site, Monroe, Wisconsin
  - Novartis Investigative Site, Neenah, Wisconsin
  - Novartis Investigative Site, Wisconsin Rapids, Wisconsin
  - Novartis Investigative Site, Casper, Wyoming
- Argentina (6):
  - Novartis Investigative Site, Jenin, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Salta
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Canada (10):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Saint John, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Guelph, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Saint Catharine's, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Novartis Investigative Site, Santiago, Chile
- Mexico (4):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Culiacan, State of Mexico
  - Novartis Investigative Site, Distrito Federal
- Puerto Rico (2):
  - Novartis Investigative Site, Guaynabo
  - Novartis Investigative Site, San Juan

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17906